CLINICAL TRIAL: NCT05983991
Title: GATA-2 Project: Retrospective and Prospective Exploratory Study for Characterisation of Predictive Parameters of Clonal Evolution in Subjects With GATA2 Germline Mutation
Brief Title: Study for Characterisation of Predictive Parameters of Clonal Evolution in Subjects With GATA2 Germline Mutation
Acronym: GATA-2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 22 HEMA 21
Record Dates: First submitted 2023-07-31; First posted 2023-08-09 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-06

CONDITIONS: GATA2 Gene Mutation
Keywords: GATA2 Gene Mutation; Myelodysplastic Syndromes; Acute myeloid Leukemia; Spectrum 2
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject with a germline GATA2 mutation (Interventional prospective cohort) (Experimental)
  Interventions: Other: Biological samples (blood and bone marrow samples).

INTERVENTIONS:
Other: Biological samples (blood and bone marrow samples). — For each included patient, biological samples (blood and bone marrow samples) will be collected at baseline visit and then during 5 years, according to the samples taken in the standard practice. No additional sampling will be performed for the study.

SUMMARY:
This trial is a translational, open-label, multi-site, retrospective and prospective cohort study of 250 patients aiming to characterize predictive parameters of clonal evolution in a population of subjects carrying the germline GATA2 mutation.

This study will be conducted on a population of subjects either with previous germline GATA2 mutation identified or newly identified for germline GATA2 mutation in the context of routine care.

Prospective cohort:

150 subjects will be included in this interventional prospective cohort study:

* Alive subjects previously identified with a germline GATA2 mutation through the already existing "Neutropenia database";
* Subject identified in the investigating centers in the context of a newly identified germline GATA2 mutation.

For each included patient, biological samples (blood and bone marrow samples) will be collected at baseline visit and then during 5 years, according to the samples taken in the standard practice. No additional sampling will be performed for the study.

Retrospective cohort:

Subjects (100 cases in total) previously identified with germline GATA2 mutation through the already existing "Neutropenia database" and with the following features may enter the retrospective cohort:

* Deceased patients,
* Lost to follow-up patients. Clinical follow-up data will be obtained from this database and/or patient's medical report.

For each retrospective case, archived blood and bone marrow samples (collected in a sanitary setting) will be sent to sponsor's centralized unit for analysis.

ELIGIBILITY:
Inclusion Criteria:

1. All subject, at any age, with a germline GATA2 mutation.
2. Patient followed in the center within a standard of care procedure or clinical trial.
3. Signed written informed consent. For minor patients: patient assent and legal guardian(s) written informed consent obtained before inclusion in the study and prior performance of any study-related procedure.
4. For French patients: patient affiliated to a Social Health Insurance.

Exclusion Criteria:

1. GATA2 somatic mutation.
2. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure.
3. Person who has forfeited his/her freedom by administrative or legal award or who is under legal protection, with the exception of persons under curatorship who may be included in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-12-07 (Actual); Primary Completion 2033-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Time to appearance of spectrum 2, defined as the delay between date of birth and appearance of an event classified as spectrum 2. | 5 years for each patient
  Spectrum 2 corresponds to MDS (Myelodysplastic Syndromes) with excess blasts, AML (Acute myeloid Leukemia) or CMML (Chronic myelomonocytic leukemia).

SECONDARY OUTCOMES:
Time to appearance of spectrum 1, defined as the delay between date of birth and appearance of spectrum 1. | 5 years for each patient
  Spectrum 1 corresponds to hypoplastic marrow and/or low-grade MDS (without excess blasts).
Time to appearance of first hematological event defined by the delay between date of birth and appearance of first hematological. | 5 years for each patient
Disease Free Survival (DFS) defined as the time from Leukemia diagnosis until first /relapse or death from any cause. | 5 years for each patient

CONTACTS AND LOCATIONS:
Locations (23):
- France (23):
  - CHU Angers, Angers
  - CHU Bordeaux, Bordeaux
  - CHU Estaing, Clermont-Ferrand
  - CHU Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - CHRU - Lille, Lille
  - IHOP Lyon, Lyon
  - CHU La Timone, Marseille
  - CHU Arnaud de Villeneuve, Montpellier
  - CHU Nantes, Nantes
  - CHU de Nice, Nice
  - Hôpital Armand Trousseau, Paris
  - Hôpital Robert Debré, Paris
  - Hôpital Saint-Louis, Paris
  - CHU Rennes, Rennes
  - CHU Hôpitaux de Rouen - Charles Nicolle, Rouen
  - CHU Saint-Etienne, Saint-Priest-en-Jarez
  - Hôpital Necker, Sèvres
  - CHU Strasbourg, Strasbourg
  - CHU Purpan - Hôpital des Enfants, Toulouse
  - Institut Universitaire Du Cancer Toulouse - Oncopole (Iuct-O), Toulouse
  - CHRU de Tours, Tours
  - CHRU Nancy Hôpital d'enfants, Vandœuvre-lès-Nancy